CLINICAL TRIAL: NCT06654271
Title: Robotic Versus Electromagnetic Bronchoscopy for Pulmonary LesIon AssessmeNT Using Integrated Intraprocedural Imaging: the RELIANT 2 Trial
Brief Title: Robotic Versus Electromagnetic Bronchoscopy for Pulmonary LesIon AssessmeNT Using Integrated Intraprocedural Imaging
Acronym: RELIANT 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rafael Paez, Assistant Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 241103
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Pulmonary Lesion; Lung Nodule, Solitary
Keywords: Electromagnetic navigation bronchoscopy; Robotic assisted bronchoscopy; Cone beam computed tomography; Diagnostic yield
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Intervention Model Description: This study will be performed as a pragmatic, cluster randomized controlled trial with parallel group assignment.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: It is not possible to blind the bronchoscopist or the patient to the platform used for each procedure, as they are both large distinctive-appearing pieces of equipment. However, allocation will be concealed until the morning of the procedure. Thoracic pathologists and bronchoscopy schedulers will remain blinded, thus allocations will not influence scheduling of procedures or histopathological interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Robotic assisted bronchoscopy (RAB) (Active Comparator): Robotic assisted bronchoscopy with integrated cone beam computed tomography
  Interventions: Device: Robotic assisted bronchoscopy (RAB)
- Electromagnetic navigation bronchoscopy (ENB) (Active Comparator): Electromagnetic navigation bronchoscopy (ENB) with integrated digital tomosynthesis
  Interventions: Device: Electromagnetic navigation bronchoscopy (ENB)

INTERVENTIONS:
Device: Robotic assisted bronchoscopy (RAB) — Participants allocated to the robotic assisted bronchoscopy arm will undergo robotic assisted bronchoscopy with integrated cone beam computed tomography
  Arms: Robotic assisted bronchoscopy (RAB)
Device: Electromagnetic navigation bronchoscopy (ENB) — Participants allocated to the electromagnetic navigation bronchoscopy arm will undergo electromagnetic navigation bronchoscopy with integrated digital tomosynthesis
  Arms: Electromagnetic navigation bronchoscopy (ENB)

SUMMARY:
RELIANT 2 is a pragmatic randomized controlled trial. The goal of this study is to compare the diagnostic yield of robotic assisted bronchoscopy with integrated cone beam computed tomography to that of electromagnetic navigation bronchoscopy with integrated digital tomosynthesis in patients undergoing bronchoscopy to biopsy a pulmonary lesion.

DETAILED DESCRIPTION:
Pulmonary nodules are an incredibly common finding, with millions incidentally detected in the US every year. Biopsy is often needed for diagnosis. There are several technologies currently available to biopsy these lesions, including electromagnetic navigational bronchoscopy (ENB) and robotic assisted bronchoscopy (RAB). The latter is used clinically with either conventional fluoroscopy or with cone beam computed tomography (CBCT) guidance, which provides real time 3-dimensional images during the procedure. Recently, CBCT has been integrated with RAB, which allows for automatic update of the lesion location. This update is believed to increase the diagnostic yield of the procedure. Given this new upgrade, we designed this pragmatic, randomized controlled study to test the hypothesis that the diagnostic yield of RAB with integrated CBCT is superior to ENB with integrated digital tomosynthesis in patients undergoing bronchoscopic biopsy of a peripheral pulmonary lesion. Patients undergoing advanced diagnostic bronchoscopy to biopsy a lung lesion will be assigned to either the RAB or ENB based on cluster randomization. Randomization will be revealed each morning before procedures are started. Any advanced diagnostic bronchoscopy scheduled on that day will be performed with the device (RAB or ENB) allocated to that room on that day. All decisions regarding procedure tools, techniques, and patient management will be per usual care and at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at time of bronchoscopy
* Scheduled for navigational bronchoscopy for the evaluation of a pulmonary lesion

Exclusion Criteria:

* Patient declines to participate
* Patients enrolled in another trial which requires the use of one specific navigational platform

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-10-14 (Actual); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the diagnostic yield, defined as the proportion of procedures that result in acquisition of lesional tissue. | 7 days post-procedure
  Lesional tissue is defined by the presence of specific pathological findings that readily explain the presence of a pulmonary lesion. The following common pathological findings are pre-specified:
  * Malignancy
  * Specific benign pathologic findings including:
    * Organizing pneumonia
    * Frank purulence/robust neutrophilic inflammation
    * Granulomatous inflammation
    * Other specific benign findings such as hamartoma, amyloidoma or other uncommon causes of peripheral pulmonary lesions with distinctive pathological patterns as adjudicated by an expert lung pathologist.

SECONDARY OUTCOMES:
Duration of bronchoscopy (in minutes) | Duration of procedure, approximately 60 minutes
  Defined as time from the start of airway registration to the removal of the bronchoscope after completion of navigation procedures

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Paez, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (3):
- United States (3):
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be made available after de-identification.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 3 months following publication of outcomes and will remain available for at least 3 years.
Access Criteria: Data will be made available to researchers who provide a methodologically sound proposal that has been approved by the Vanderbilt Institutional Review Board and the study executive committee.

REFERENCES:
- [Background] Zhang C, Xie F, Li R, Cui N, Herth FJF, Sun J. Robotic-assisted bronchoscopy for the diagnosis of peripheral pulmonary lesions: A systematic review and meta-analysis. Thorac Cancer. 2024 Mar;15(7):505-512. doi: 10.1111/1759-7714.15229. Epub 2024 Jan 29. PMID 38286133
- [Background] Kalchiem-Dekel O, Connolly JG, Lin IH, Husta BC, Adusumilli PS, Beattie JA, Buonocore DJ, Dycoco J, Fuentes P, Jones DR, Lee RP, Park BJ, Rocco G, Chawla M, Bott MJ. Shape-Sensing Robotic-Assisted Bronchoscopy in the Diagnosis of Pulmonary Parenchymal Lesions. Chest. 2022 Feb;161(2):572-582. doi: 10.1016/j.chest.2021.07.2169. Epub 2021 Aug 9. PMID 34384789
- [Background] Low SW, Lentz RJ, Chen H, Katsis J, Aboudara MC, Whatley S, Paez R, Rickman OB, Maldonado F. Shape-Sensing Robotic-Assisted Bronchoscopy vs Digital Tomosynthesis-Corrected Electromagnetic Navigation Bronchoscopy: A Comparative Cohort Study of Diagnostic Performance. Chest. 2023 Apr;163(4):977-984. doi: 10.1016/j.chest.2022.10.019. Epub 2022 Oct 29. PMID 36441041
- [Background] Katsis J, Roller L, Aboudara M, Pannu J, Chen H, Johnson J, Lentz RJ, Rickman O, Maldonado F. Diagnostic Yield of Digital Tomosynthesis-assisted Navigational Bronchoscopy for Indeterminate Lung Nodules. J Bronchology Interv Pulmonol. 2021 Oct 1;28(4):255-261. doi: 10.1097/LBR.0000000000000766. PMID 33734149
- [Background] Gould MK, Tang T, Liu IL, Lee J, Zheng C, Danforth KN, Kosco AE, Di Fiore JL, Suh DE. Recent Trends in the Identification of Incidental Pulmonary Nodules. Am J Respir Crit Care Med. 2015 Nov 15;192(10):1208-14. doi: 10.1164/rccm.201505-0990OC. PMID 26214244
- [Background] Nadig TR, Thomas N, Nietert PJ, Lozier J, Tanner NT, Wang Memoli JS, Pastis NJ, Silvestri GA. Guided Bronchoscopy for the Evaluation of Pulmonary Lesions: An Updated Meta-analysis. Chest. 2023 Jun;163(6):1589-1598. doi: 10.1016/j.chest.2022.12.044. Epub 2023 Jan 11. PMID 36640994
- [Background] Criner GJ, Eberhardt R, Fernandez-Bussy S, Gompelmann D, Maldonado F, Patel N, Shah PL, Slebos DJ, Valipour A, Wahidi MM, Weir M, Herth FJ. Interventional Bronchoscopy. Am J Respir Crit Care Med. 2020 Jul 1;202(1):29-50. doi: 10.1164/rccm.201907-1292SO. PMID 32023078
- [Background] Agrawal A, Hogarth DK, Murgu S. Robotic bronchoscopy for pulmonary lesions: a review of existing technologies and clinical data. J Thorac Dis. 2020 Jun;12(6):3279-3286. doi: 10.21037/jtd.2020.03.35. PMID 32642251
- [Background] Aboudara M, Roller L, Rickman O, Lentz RJ, Pannu J, Chen H, Maldonado F. Improved diagnostic yield for lung nodules with digital tomosynthesis-corrected navigational bronchoscopy: Initial experience with a novel adjunct. Respirology. 2020 Feb;25(2):206-213. doi: 10.1111/resp.13609. Epub 2019 Jul 2. PMID 31265204
- [Background] Styrvoky K, Schwalk A, Pham D, Madsen K, Chiu HT, Abu-Hijleh M. Radiation dose of cone beam CT combined with shape sensing robotic assisted bronchoscopy for the evaluation of pulmonary lesions: an observational single center study. J Thorac Dis. 2023 Sep 28;15(9):4836-4848. doi: 10.21037/jtd-23-587. Epub 2023 Aug 30. PMID 37868864
- [Derived] Paez R, Ratwani AP, Duke JD, Bridwell G, Leonard K, Katsis JM, Pickering EM, Thiboutot J, Chen H, Chen SC, Shojaee S, Yarmus L, Lentz RJ, Maldonado F; Interventional Pulmonary Outcomes Group. Robotic versus electromagnetic bronchoscopy for pulmonary leslon assessment using integrated intraprocedural imaging: Study protocol for the reliant 2 trial. PLoS One. 2025 Dec 3;20(12):e0327611. doi: 10.1371/journal.pone.0327611. eCollection 2025. PMID 41336287
- [Derived] Chen SC, Chen H, Paez R, Gatto CL, Lentz RJ, Maldonado F. A randomization strategy for a cluster-randomized controlled trial with variable operating room availability. Contemp Clin Trials. 2025 Oct;157:108057. doi: 10.1016/j.cct.2025.108057. Epub 2025 Aug 28. PMID 40885487